CLINICAL TRIAL: NCT01432457
Title: A Phase IV, Multicenter, Randomized, 8-Week, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy of 2 Fixed Doses (50 and 100 mg/Day) of Desvenlafaxine Succinate Sustained-Release (DVS SR) in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained-Release (DVS SR) in Adult Outpatients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2061028; 3151A1-4420
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- desvenlafaxine succinate sustained-release 50 mg/day (Experimental)
  Interventions: Drug: desvenlafaxine succinate sustained-release 50 mg/day
- desvenlafaxine succinate sustained-release 100 mg/day (Experimental)
  Interventions: Drug: desvenlafaxine succinate sustained-release 100 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained-release 50 mg/day — 50 mg tablets of DVS SR taken orally once daily for 8 weeks; 1 week of placebo taper
  Other Names: Pristiq
  Arms: desvenlafaxine succinate sustained-release 50 mg/day
Drug: desvenlafaxine succinate sustained-release 100 mg/day — 100 mg tablets of DVS SR taken orally once daily for 8 weeks (which includes 1 week of titration at 50 mg/day); 1 week of taper at 50 mg/day
  Arms: desvenlafaxine succinate sustained-release 100 mg/day
Drug: placebo — 50 mg and 100 mg placebo matching tablets taken orally once daily for 8 weeks; 1 week of placebo taper
  Arms: Placebo

SUMMARY:
A multicenter, 8-week study to evaluate the efficacy of 2 doses (50 and 100 mg/day) of desvenlafaxine succinate sustained-release (DVS SR) versus placebo in adult outpatients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 years or older who are fluent in written and spoken English.
* A primary diagnosis of MDD based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM- IV-TR), single or recurrent episode, without psychotic features.
* A HAM-D17 total score ≥20 at the screening and baseline (study day -1) visits and no more than a 4-point improvement from screening to baseline.

Exclusion Criteria:

* Significant risk of suicide based on clinical judgment.
* Current (within 12 months before baseline) psychoactive substance abuse or dependence (including alcohol), manic episode, posttraumatic stress disorder, obsessive compulsive disorder, or a lifetime diagnosis of bipolar or psychotic disorder.
* Current generalized anxiety disorder, panic disorder, or social anxiety disorder.
* History or current evidence of gastrointestinal disease known to interfere with the absorption or excretion of drugs or a history of surgery known to interfere with the absorption or excretion of drugs.
* Any unstable hepatic, renal, pulmonary, cardiovascular, ophthalmologic, neurologic, or other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (61):
- United States (61):
  - Dedicated Clinical Research, Phoenix, Arizona
  - Deidcated Clinical Research, Phoenix, Arizona
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Southwestern Research, Incorporated, Beverly Hills, California
  - Clinical Innovations, Inc., Costa Mesa, California
  - Synergy Clinical Research of Escondido, Escondido, California
  - Synergy Clinical Research Center, National City, California
  - Pacific Research Partners, Oakland, California
  - Pasadena Research Institute, LLC, Pasadena, California
  - Clinical Innovations, Inc., Riverside, California
  - Affiliated Research Institute, San Diego, California
  - Clinical Innovations, Inc., San Diego, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Viking Clinical Research Center, Temecula, California
  - Collaborative Neuroscience Network, Inc. South Bay, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Clinical Neuroscience Solutions Incorporated, Jacksonville, Florida
  - Accurate Clinical Trials, Inc., Kissimmee, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Comprehensive NeuroScience, Incorporated, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR-Baber Research Inc., Naperville, Illinois
  - American Medical Research, Inc., Oak Brook, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Via Christi Research, Wichita, Kansas
  - Pharmasite Research Inc, Baltimore, Maryland
  - Midwest Research Group, Saint Charles, Missouri
  - Heartland Pharma Development, North Platte, Nebraska
  - CRI Worldwide, LLC, Marlton, New Jersey
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Medical and Behavioral Health Research Pc, New York, New York
  - Prairie St. Johns Clinic - Fargo, Fargo, North Dakota
  - Odyssey Research, Fargo, North Dakota
  - Plains Medical Clinic, Fargo, North Dakota
  - NorthCoast Clinical Trials Inc., Beachwood, Ohio
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Carolina Clinical Research Services, Columbia, South Carolina
  - FutureSearch Trials, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Radiant Research, Inc., Murray, Utah
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Clayton AH, Tourian KA, Focht K, Hwang E, Cheng RF, Thase ME. Desvenlafaxine 50 and 100 mg/d versus placebo for the treatment of major depressive disorder: a phase 4, randomized controlled trial. J Clin Psychiatry. 2015 May;76(5):562-9. doi: 10.4088/JCP.13m08978. PMID 25375652
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061028&StudyName=Study%20Evaluating%20Desvenlafaxine%20Succinate%20Sustained-Release%20%28DVS%20SR%29%20in%20Adult%20Outpatients%20with%20Major%20Depressive%20Disorder%20%28MDD%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the United States from October 2011 to May 2012.
Pre-assignment Details: Subjects were screened up to 2 weeks.
Groups:
- Placebo: Placebo group received placebo tablets through 8-weeks of double-blind treatment and during 1-week of taper.
- DVS SR 50 mg: Desvenlafaxine Succinate Sustained Release (DVS SR) 50 milligrams (mg) group received 50 mg DVS SR tablets through the 8-weeks of double-blind treatment and received placebo tablets each day during 1-week taper.
- DVS SR 100 mg: Desvenlafaxine Succinate Sustained Release (DVS SR) 100 milligrams (mg) group received 50 mg DVS SR tablets each day for first week of treatment, 100 mg DVS SR tablets each day through the remainder of the 8-week double-blind treatment and received 50 mg DVS SR tablets each day during 1-week taper.
Period: Overall Study
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Started | 306 | 306 | 312
Completed | 269 | 258 | 253
Not Completed | 37 | 48 | 59
Not completed — Adverse Event | 7 | 10 | 16
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Lost to Follow-up | 11 | 15 | 20
Not completed — Protocol Violation | 3 | 2 | 6
Not completed — Withdrawal by Subject | 6 | 11 | 9
Not completed — Reasons not defined | 2 | 3 | 4
Not completed — Did not take study drug | 6 | 6 | 3

BASELINE CHARACTERISTICS:
Population: The numbers are correct. Participants flow starts with all randomized subjects while baseline is summarized for safety population defined as randomized AND took at least one dose. Started- (Other Did not take study drug) is the number for baseline summary.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg | Total
Number analyzed (Participants) | 300 | 300 | 309 | 909
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.72 (12.42) | 41.78 (13.56) | 41.30 (12.80) | 41.60 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 172 | 165 | 510
  Male | 127 | 128 | 144 | 399

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Hamilton Rating Scale for Depression, 17-item Total Score (HAM-D17) at Week 8
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Each item is scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), for a maximum total score of 52; higher scores indicate more depression. Change from baseline: score at observation minus score at baseline.
Time Frame: Baseline to Week 8 (final on-therapy)
Population: Intent-To-Treat (ITT) population: randomized subjects who have taken at least 1 dose of double-blind investigational product, and had a baseline and at least 1 post-baseline HAM-D17 total score. Imputation technique: A mixed effects model for repeated measures (MMRM) was used with the baseline HAM-D17 score as a covariate.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 267 | 257 | 252
Units on a scale | -9.71 (0.42) | -11.28 (0.42) | -11.67 (0.42)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; A mixed effects model for repeated measures (MMRM) with treatment, visit, treatment by visit interaction, and site as fixed effects, and the baseline HAM-D17 score as a covariate was used to compare DVS SR dose to placebo. The test of the null hypothesis was used study-wise with alpha = 0.05 (2-sided); Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — A Hochberg step-up procedure was used to control for the multiplicity associated with multiple active dose arms; Adjusted Mean Difference = 1.57, 95% CI 2-sided [0.44 to 2.69]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A Hochberg step-up procedure was used to control for the multiplicity associated with multiple active dose arms; Adjusted Mean Difference = 1.96, 95% CI 2-sided [0.84 to 3.08]

2. Primary Outcome: Change From Baseline on the Hamilton Rating Scale for Depression, 17-item Total Score (HAM-D17) at Week 8
Description: as for outcome 1
Time Frame: Baseline to Week 8 (final on-therapy)
Population: Intent-To-Treat (ITT) population: randomized subjects who have taken at least 1 dose of double-blind investigational product, and had a baseline and at least 1 post-baseline HAM-D17 total score. Imputation technique: Analysis of covariance (ANCOVA) was used based on last-observation-carried-forward (LOCF) data.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 294 | 291 | 301
Units on a scale | -9.50 (0.44) | -10.86 (0.43) | -11.16 (0.43)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; To assess the sensitivity of the results to the missing data assumptions, an analysis of covariance (ANCOVA) model based on the last observation carried forward (LOCF) was used. The test of the null hypothesis was used study-wise with alpha = 0.05 (2-sided); Test type: Superiority or Other; p = 0.014, ANCOVA; Adjusted Mean Difference = 1.36, 95% CI 2-sided [0.28 to 2.45]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA; Adjusted Mean Difference = 1.67, 95% CI 2-sided [0.59 to 2.74]

3. Secondary Outcome: Change From Baseline on the Clinical Global Impression Scale-Improvement (CGI-I)
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Higher score = worse outcome.
Time Frame: Baseline to Week 8 (final on-therapy)
Population: Intent-To-Treat (ITT) population: randomized subjects who have taken at least 1 dose of double-blind investigational product, and had a baseline and at least 1 post-baseline HAM-D17 total score. Imputation technique: The Cochran-Mantel-Haenszel row-mean-score-difference test using ridit scores based on last-observation-carried-forward (LOCF) data.
Measure: Number; unit: number of participants
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 294 | 291 | 301
number of participants
  1=Very much improved | 55 | 57 | 81
  2=Much improved | 76 | 104 | 98
  3=Minimally improved | 83 | 79 | 69
  4=No change | 73 | 48 | 49
  5=Minimally worse | 7 | 3 | 4
  6=Much worse | 0 | 0 | 0
  7=Very much worse | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; CGI-I was analyzed with the Cochran-Mantel-Haenszel row-mean-score-difference test using ridit scores. Each DVS SR arm was separately compared to placebo controlling for site. The test of the null hypothesis was used study-wise with alpha = 0.05 (2-sided); Test type: Superiority or Other; p = 0.029, Cochran-Mantel-Haenszel — p-value was obtained from the separate pair-wise Cochran-Mantel-Haenszel test versus placebo for the alternative hypothesis of "Row Mean Scores Differences" controlling for site
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline on the Clinical Global Impression-Severity Score (CGI-S)
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = worse state.
Time Frame: Baseline to Week 8 (final on-therapy)
Population: Intent-To-Treat (ITT) population: randomized subjects who have taken at least 1 dose of double-blind investigational product, and had a baseline and at least 1 post-baseline HAM-D17 total score. Imputation technique: A mixed effects model for repeated measures (MMRM) was used with the baseline CGI-S score as a covariate.
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 265 | 257 | 252
Units on scale | -1.27 (0.06) | -1.47 (0.06) | -1.55 (0.06)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; CGI-S was analyzed using the mixed effects model for repeated measures (MMRM) with treatment, visit, treatment by visit interaction, and site as fixed effects, and the baseline CGI-S score as a covariate. The test of the null hypothesis was used study-wise with alpha = 0.05 (2-sided); Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; Adjusted Mean Difference = 0.20, 95% CI 2-sided [0.05 to 0.34]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = 0.28, 95% CI 2-sided [0.13 to 0.43]

5. Secondary Outcome: Change From Baseline on the Clinical Global Impression-Severity (CGI-S) Score
Description: as for outcome 4
Time Frame: Baseline to Week 8 (final on-therapy)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 294 | 291 | 301
Units on scale | -1.21 (0.07) | -1.38 (0.07) | -1.43 (0.07)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.062, ANCOVA; Adjusted Mean Difference = 0.17, 95% CI 2-sided [-0.01 to 0.34]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.014, ANCOVA; Adjusted Mean Difference = 0.22, 95% CI 2-sided [0.04 to 0.39]

6. Secondary Outcome: Hamilton Rating Scale for Depression, 17-item (HAM-D17) Response Rate
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Each item is scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), for a maximum total score of 52; higher scores indicate more depression. A response is defined as ≥ 50% decrease from baseline on Hamilton Psychiatric Rating Scale for Depression (HAM-D17) total score.
Time Frame: Baseline to Week 8 (final on-therapy)
Population: Intent-to-Treat (ITT) population: randomized subjects who have taken at least 1 dose of double-blind investigational product, and had a baseline and at least one post-baseline HAM-D17 total score. Imputation technique: A logistic regression model based on last-observation-carried-forward (LOCF) data was used.
Measure: Number; unit: percentage of the number of participants
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 294 | 291 | 301
percentage of the number of participants | 39.46 | 45.02 | 47.51
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Response in HAM-D17 was analyzed based on a logistic regression model with treatment and site as fixed factors and the baseline HAM-D17 total score as a covariate. The test of the null hypothesis was used study-wise with alpha = 0.05 (2-sided); Test type: Superiority or Other; p = 0.198, Regression, Logistic; Adjusted Odds Ratio = 1.242, 95% CI 2-sided [0.893 to 1.726]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.054, Regression, Logistic; Adjusted Odds Ratio = 1.378, 95% CI 2-sided [0.995 to 1.910]

7. Secondary Outcome: Hamilton Rating Scale for Depression, 17-item (HAM-D17) Remission Rate
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Each item is scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), for a maximum total score of 52; higher scores indicate more depression. Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) total score of ≤ 7.
Time Frame: Baseline to week 8 (final on-therapy)
Population: Intent-to-Treat (ITT) population: randomized subjects who have taken at least 1 dose of double-blind investigational product, and had a baseline and at least one post-baseline HAM-D17 total score. Imputation technique: A logistic regression model based on last- observation-carried-forward (LOCF) data was used.
Measure: Number; unit: percentage of the number of participants
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 294 | 291 | 301
percentage of the number of participants | 21.77 | 24.05 | 28.57
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; Remission in HAM-D17 was analyzed based on a logistic regression model with treatment and site as fixed factors and the baseline HAM-D17 total score as a covariate. The test of the null hypothesis was used study-wise with alpha = 0.05 (2-sided); Test type: Superiority or Other; p = 0.615, Regression, Logistic; Adjusted Odds Ratio = 1.105, 95% CI 2-sided [0.749 to 1.631]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.072, Regression, Logistic; Adjusted Odds Ratio = 1.412, 95% CI 2-sided [0.969 to 2.057]

8. Secondary Outcome: Change From Baseline on the Arizona Sexual Experiences (ASEX) Scale Total Score
Description: The ASEX scale has 5 items to assess sexual functioning with a 1-week recall period. The 5 items assess sex drive, ease of arousal, ease of erection/lubrication, ease of orgasm and orgasm satisfaction. Subjects were encouraged to complete all 5 items regardless of sexual activity during the past week. However, all analyses utilized only the data for the visits where the presence of sexual activity was indicated.
  Each individual score ranged from 1 to 6; the total score (based on the sum of the individual items) ranged from 5 to 30; higher scores indicated worse sexual function.
Time Frame: Baseline to Week 8 (final on-therapy)
Population: Safety population: randomized subjects who have taken at least 1 dose of double-blind investigational product. Imputation technique: ASEX scale total score analyzed using analysis of covariance based on LOCF data. ASEX data only analyzed for subjects indicating sexual activity at baseline and a timepoint during post-baseline.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Number analyzed (Participants) | 135 | 138 | 149
Units on a scale | -0.45 (0.36) | -0.35 (0.35) | -0.13 (0.33)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 50 mg; The treatment by gender interaction was first tested using an analysis of covariance (ANCOVA) model with treatment, site, gender, and treatment by gender as factors and the baseline total score as a covariate. The test of the null hypothesis was used study-wise with alpha = 0.05 (2-sided); Test type: Superiority or Other; p = 0.837, ANCOVA — p-value was obtained from the ANCOVA model as change from baseline = Treatment + Site + Gender + Baseline; Adjusted Mean Difference = -0.09, 95% CI 2-sided [-0.98 to 0.80]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 100 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.471, ANCOVA — p-value was obtained from the ANCOVA model as change from baseline = Treatment + Site + Gender + Baseline; Adjusted Mean Difference = -0.32, 95% CI 2-sided [-1.19 to 0.55]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | DVS SR 50 mg | DVS SR 100 mg
Serious Adverse Events (participants affected / at risk) | 6/300 | 2/300 | 2/309
Other Adverse Events (participants affected / at risk) | 110/300 | 159/300 | 163/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=300) | DVS SR 50 mg (N=300) | DVS SR 100 mg (N=309)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Serum serotonin increased (Investigations) | 0 | 1 | 0 — Significantly elevated serotonin level
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 — Abnormal behavior as a result of reaction to alcohol and unknown substance
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0 — Increased depressive symptoms
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=300) | DVS SR 50 mg (N=300) | DVS SR 100 mg (N=309)
Constipation (Gastrointestinal disorders) | 11 | 17 | 12
Diarrhoea (Gastrointestinal disorders) | 18 | 26 | 19
Dry mouth (Gastrointestinal disorders) | 24 | 31 | 37
Nausea (Gastrointestinal disorders) | 24 | 48 | 52
Fatigue (General disorders) | 7 | 10 | 17
Decreased appetite (Metabolism and nutrition disorders) | 5 | 12 | 18
Dizziness (Nervous system disorders) | 14 | 28 | 32
Headache (Nervous system disorders) | 32 | 57 | 61
Somnolence (Nervous system disorders) | 12 | 17 | 16
Insomnia (Psychiatric disorders) | 11 | 20 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.